CLINICAL TRIAL: NCT00512096
Title: A Phase II Study of (Neoadjuvant Chemotherapy Trial Prior to Extirpative Surgery) for Clinical Stage TanyN2-3M0 Squamous Cell Carcinoma of the Penis
Brief Title: Neoadjuvant Chemotherapy for Patients With Squamous Cell Carcinoma of the Penis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-194
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Penile Cancer
Keywords: Genitourinary; Penile Cancer; Neoadjuvant Chemotherapy; Extirpative Surgery; TanyN2-3M0 Squamous Cell Carcinoma of the Penis; Cisplatin; Platinol-AQ; Platinol; CDDP; Ifosfamide; Ifex; Paclitaxel; Taxol
MeSH Terms: conditions — Penile Neoplasms | interventions — Ifosfamide; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin + Ifosfamide + Paclitaxel (Experimental): Cisplatin 25 mg/m^2 IV Days 1-3; Ifosfamide 1200 mg/m^2 IV Days 1-3; Paclitaxel 175 mg/m^2 IV Day 1
  Interventions: Drug: Ifosfamide; Drug: Paclitaxel (Taxol); Drug: Cisplatin

INTERVENTIONS:
Drug: Ifosfamide — 1200 mg/m^2 By Vein Over 2 Hours on Days 1-3
  Other Names: Ifex
Drug: Paclitaxel (Taxol) — 175 mg/m^2 By Vein Over 3 Hours on Day 1
  Other Names: Taxol
Drug: Cisplatin — 25 mg/m^2 By Vein Over 2 Hours on Days 1-3
  Other Names: Platinol-AQ; Platinol; CDDP

SUMMARY:
Primary Objective:

-To evaluate the feasibility and efficacy of multimodality treatment (neoadjuvant chemotherapy prior to extirpative surgery) for clinical stage TXN2-3M0 squamous cell carcinoma of the penis.

DETAILED DESCRIPTION:
Before treatment starts, participants will have a complete exam, including blood and urine tests. A CT scan of the abdomen and pelvis will be done. Participants will have a chest x-ray, bone scan, and an EKG (heart test). A special heart function test may also need to be done in some participants. If necessary a biopsy of enlarged lymph node(s) will be obtained prior to treatment.

Blood tests will be repeated once a week during treatment. CT scans of the abdomen and pelvis and a Chest x-ray will be done after 2 treatments with Taxol, Ifosfamide, and Cisplatin. These will also be done before surgery.

The drugs Taxol, Ifosfamide and Cisplatin will be given through a catheter (plastic tube) placed in a vein in the arm or under the collarbone. Taxol will be given over 3 hours the first day of the treatment cycle. To prevent an allergic reaction, before the Taxol is given, the participant will receive three drugs. These are Dexamethasone, Diphenhydramine, and either Cimetidine or Ranitidine.

After Taxol, Ifosfamide will be given over 2 hours every day for the first three days of the treatment cycle. To prevent possible irritation of Ifosfamide to the bladder, participants will also receive Mesna through the plastic catheter. Mesna will be given both before and after Ifosfamide every day. Mesna is not chemotherapy. It is a medication to prevent side effects of Ifosfamide into the bladder.

Every day for the first three days of the cycle, and after Ifosfamide is given, participants will also receive Cisplatin through the catheter at a steady rate over 2 hours, along with Mannitol and salt water to flush the kidneys. This treatment will be given in the hospital and will require staying in the hospital for 3-4 days. It will be repeated for a total of 4 times; once every 21 days, if the participant has high enough numbers of white blood cells and platelets.

Participants may be given injections of G-CSF under the skin once a day for up to 7 days (days 6-12 of the cycle) to bring the white cells up faster after the chemotherapy. This will also lower the risk of severe infections.

After completing 4 treatments of chemotherapy, participants will have blood and urine tests, a chest x-ray to learn the response of the tumor to the chemotherapy. They will also have a CT scan of the abdomen and pelvis. Participants who have a response to the chemotherapy, or show no sign of new spread of the cancer to other parts of the body, will then have surgery. Surgery will be done to remove the tumor. The lymph nodes in the groin will be removed. The pelvic lymph nodes may also need to be removed. How much tissue is removed depends on how far the tumor has spread. The surgeons will explain the specifics of the surgery in a separate consent form.

After completion of the treatment, physical exams, CT scans, chest x-rays, blood tests, and urine tests will be done every 3 months for 2 years. They will then be done every 6 months. These procedures can be done by a physician at M. D. Anderson or by the participant's own doctor. If the participant's doctor does it, the information will need to be forwarded to the doctors at M. D. Anderson. Participants will be expected to come to M. D. Anderson or to their respective participating urologist/medical oncologist at least once every 6 months for a check-up.

This is an investigational study. The FDA has approved Taxol, Ifosfamide, Cisplatin, and Mesna. Up to 40 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from each patient prior to study entry.
2. Age >/= 14 years of age. Life expectancy greater than or equal to 6 months. PS </= 2 (ECOG).
3. Patients with histologically confirmed squamous cell carcinoma of the penis who present with clinical stage (T(subscript)xN(subscript)2-3M(subscript)0) disease based on the 1987-1992 TNM Staging System and meeting the additional clinicopathologic criteria as defined in the protocol (section 3.1).
4. Patients must have adequate physiologic reserve as evidenced by: absolute neutrophil count (ANC) >/= 1,500/mm3(superscript) and platelet count >/= 100,000/mm3. Transaminases </= 2 times the upper limit of normal. Conjugated bilirubin </= 1.5mg/dL. Creatinine clearance (either calculated or measured) of >/= 40ml/minute.
5. No evidence of active ischemia on the EKG and, for patients with significant prior coronary artery disease history, an ejection fraction of more than 40%. No evidence of severe conduction abnormalities on EKG.

Exclusion Criteria:

1. Patients with uncontrolled infection or CNS disease.
2. Distant metastasis (TNM stage M1, i.e., lung, bone, other visceral sites, lymph node metastasis above the aortic bifurcation).
3. Patients with clinically negative inguinal examinations or those with palpable adenopathy not meeting pathological or clinical criteria (i.e., minimal nodal metastasis or false positive inguinal examination).
4. Prior systemic chemotherapy for penile carcinoma.
5. Prior radiation therapy to inguinal or pelvic lymph nodes.

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Pagliaro LC, Williams DL, Daliani D, Williams MB, Osai W, Kincaid M, Wen S, Thall PF, Pettaway CA. Neoadjuvant paclitaxel, ifosfamide, and cisplatin chemotherapy for metastatic penile cancer: a phase II study. J Clin Oncol. 2010 Aug 20;28(24):3851-7. doi: 10.1200/JCO.2010.29.5477. Epub 2010 Jul 12. PMID 20625118
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 17-AUG-99 to 15-OCT-08; all participants were recruited at MD Anderson Cancer Center
Period: Overall Study
Arm/Group | Cisplatin + Ifosfamide + Paclitaxel
Started | 30
Completed | 23
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin + Ifosfamide + Paclitaxel
Number analyzed (Participants) | 30
Age Continuous [Median (Full Range); unit: years] | 57.5 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Remission (pCR)
Description: Histopathologic assessment of surgical resection to confirm Pathologoic Complete Remission. Complete remission defined as disappearance of all target lesions.
Time Frame: restaging with second and fourth 21-day cycles followed by surgery
Population: Participants who completed chemotherapy without progression then had surgical resection.
Measure: Number; unit: participants
Arm/Group | Cisplatin + Ifosfamide + Paclitaxel
Number analyzed (Participants) | 30
participants | 3

ADVERSE EVENTS:
Time Frame: Nine years and 6 months
Arm/Group | Cisplatin + Ifosfamide + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 13/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cisplatin + Ifosfamide + Paclitaxel (N=30)
allergic reaction (Immune system disorders) | 1/23 (1)
myocarcial ischemia (Cardiac disorders) | 2/23 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin + Ifosfamide + Paclitaxel (N=30)
anemia (Blood and lymphatic system disorders) | 1 (1) — grade 3 only, no grade 4 events
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — grade 4 only, no grade 3 events
infection (Infections and infestations) | 5 (5) — grade 3 events, no grade 4
deep vein thrombosis (Vascular disorders) | 1 (1) — no grade 4 events
central venous catheter related thrombosis (Vascular disorders) | 1 (1) — grade 3, no grade 4 events
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — grade 3, no grade 4 events
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — grade 3 event, no grade 4 events
neuropathy motor (Nervous system disorders) | 1 (1) — grade 3 event, no grade 4 events
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — grade 3 event, no grade 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No